CLINICAL TRIAL: NCT04921098
Title: Evaluation of Diode Laser Cyclophotocoagulation in Adult Refractory Glaucoma
Brief Title: CPC in Adult Refractory Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mina Abdelmalek Besada, Principal Investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-05-01
Record Dates: First submitted 2021-05-30; First posted 2021-06-10 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Refractory Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Refractory glaucoma (Experimental)
  Interventions: Procedure: Diode Laser Cyclophotocoagulation

INTERVENTIONS:
Procedure: Diode Laser Cyclophotocoagulation — A handpiece (G probe) is used to deliver the diode laser energy with a wavelength of 810 nm.

SUMMARY:
The purpose of this study is to assess the relative effectiveness and safety of diode laser cyclophotocoagulation procedure to reduce IOP and relieve pain in adult patients with refractory glaucoma.

DETAILED DESCRIPTION:
A hospital -based, prospective interventional non comparative case series study.This study will be conducted on patients with refractory glaucoma whose ages are 18 years and older.They will be subjected to Transscleral Diode Laser Cyclophotocoagulation.

Postoperative evaluation will be scheduled for the first day postoperative, then 1 week later and then at 1st, 3rd, month postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Patients with refractory glaucoma aging 18 years and older.
  2. Both sexes are included.
  3. Patients Capable of giving informed consent.
  4. Pseudophkic glaucoma.
  5. Aphakic glaucoma.
  6. Silicon oil induced glaucoma.
  7. Neovascular glaucoma.
  8. Inflammatory glaucoma.

Exclusion Criteria:

1. Patients <18 years of age.
2. Patients controlled on regular antiglaucomatous therapy.
3. Patients who cannot do regular follow up visits.
4. Diffuse scleral staphyloma at the site of CPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
change in intraocular pressure | First day postoperative and 1 week
  IOP measuring using Goldmann applanation tonometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

REFERENCES:
- [Background] Ansari E, Gandhewar J. Long-term efficacy and visual acuity following transscleral diode laser photocoagulation in cases of refractory and non-refractory glaucoma. Eye (Lond). 2007 Jul;21(7):936-40. doi: 10.1038/sj.eye.6702345. Epub 2006 Apr 21. PMID 16628239
- [Background] Lai JS, Tham CC, Chan JC, Lam DS. Diode laser transscleral cyclophotocoagulation in the treatment of chronic angle-closure glaucoma: a preliminary study. J Glaucoma. 2003 Aug;12(4):360-4. doi: 10.1097/00061198-200308000-00011. PMID 12897582
- [Background] Nassiri N, Kamali G, Rahnavardi M, Mohammadi B, Nassiri S, Rahmani L, Nassiri N. Ahmed glaucoma valve and single-plate Molteno implants in treatment of refractory glaucoma: a comparative study. Am J Ophthalmol. 2010 Jun;149(6):893-902. doi: 10.1016/j.ajo.2010.01.025. Epub 2010 May 8. PMID 20451896